CLINICAL TRIAL: NCT02860884
Title: Using Infrared Spectroscopy for Diagnosis Severity of Nonalcoholic Fatty Liver Disease
Acronym: NASH
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC13_8989
Record Dates: First submitted 2016-07-26; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Fatty Liver; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- simple fatty liver: patients with fatty liver disease
  Interventions: Procedure: liver biopsy; Other: infrared spectroscopy
- NASH: patients with nonalcoholic steatohepatitis
  Interventions: Procedure: liver biopsy; Other: infrared spectroscopy

INTERVENTIONS:
Procedure: liver biopsy
Other: infrared spectroscopy

SUMMARY:
The main objective of this study is to evaluate the ability of infrared spectroscopy to discriminate simple hepatic steatosis from NASH

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a liver biopsy for simple fatty liver or NASH and for which a serum sample is serum bank
* Men or Women
* aged of 18 years or more
* After giving their consent to participate in research

Exclusion Criteria:

* Known Cancer
* Refusal of consent
* Inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a liver biopsy for simple fatty liver or NASH and for which a serum sample is serum bank
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity | through study completion, an average of 1 year
  Evaluation of the ability of infrared spectroscopy to discriminate simple hepatic steatosis from NASH with liver biopsy as a gold standard

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No